CLINICAL TRIAL: NCT03871166
Title: Hemoglobin Concentration in Patients With an Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan Adriaan Graw, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: RECETTA
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood transfusion — Observational post-ad-hoc design to compare patients admitted with an ARDS and separated into different groups according to their mean hemoglobin concentration during their stay on the intensive care unit.
  Approximately 1000 adult patients admitted from 2007 to 2018 to the Charite ARDS center will be enrolled in the study. They are followed up until their discharge from the ICU.
  [Time Frame: 01/2007 - 12/2018]

SUMMARY:
Retrospective analysis of hemoglobin concentrations and red cell transfusion thresholds in patients with an Acute Respiratory Distress Syndrome (ARDS) admitted to an ARDS-center of a German university hospital.

DETAILED DESCRIPTION:
Transfusion of packed red blood cells is a common procedure in critically ill patients. In recent years it has been shown that for many patient populations a restrictive transfusion strategy is not inferior compared to a liberal transfusion strategy with regard to overall outcome.

So far it is unclear whether patients with an ARDS should receive blood transfusions according to a restrictive or liberal transfusion strategy. Besides pulmonary gar exchange and cardiac output, the hemoglobin concentration is an important determinant for oxygen delivery.

The aim of this retrospective observational study is to analyze if low levels of hemoglobin/a restrictive transfusion strategy and are associated with a different mortality compared to higher levels of hemoglobin/a liberal transfusion strategy in patients with an ARDS.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with ARDS
* Admission to the Charité ARDS center

Exclusion Criteria:

* All patients <18 years at the time of admission
* All patients with ARDS not admitted to the Charité ARDS center

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with ARDS and admitted to the ICUs of the Charité ARDS center will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 01/2007 - 12/2018
  Mortality of patients with ARDS at 28 days according to transfusion threshold

SECONDARY OUTCOMES:
Failure-free days composites | 01/2007 - 12/2018
  Failure-free days composites according to transfusion threshold

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Graw, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Campus Virchow-Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Hunsicker O, Materne L, Bunger V, Krannich A, Balzer F, Spies C, Francis RC, Weber-Carstens S, Menk M, Graw JA. Lower versus higher hemoglobin threshold for transfusion in ARDS patients with and without ECMO. Crit Care. 2020 Dec 16;24(1):697. doi: 10.1186/s13054-020-03405-4. PMID 33327953